CLINICAL TRIAL: NCT02374333
Title: Pilot Study of Redirected Autologous T Cells Engineered to Contain Humanized Anti-CD19 Attached to TCRζ and 4-1BB Signaling Domains in Patients With Relapsed or Refractory CD19+ Leukemia and Lymphoma Previously Treated With Cell Therapy
Brief Title: Pilot Study of Redirected Autologous T Cells Engineered to Contain Humanized Anti-CD19 in Patients With Relapsed or Refractory CD19+ Leukemia and Lymphoma Previously Treated With Cell Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13BT022, 819851
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Acute Lymphocytic Leukemia; Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- huCART19 (Experimental): CART19 cells transduced with a lentiviral vector to express humanized anti-CD19 administered by IV injection
  Interventions: Biological: huCART19

INTERVENTIONS:
Biological: huCART19
  Other Names: huCTL019

SUMMARY:
This is a pilot study to evaluate humanized CD19 redirected autologous T cells (or huCART19 cells) in patients with relapsed or refractory CD19+ leukemia and lymphoma that was previously treated with cell therapy. This study is targeting pediatric patients aged 1-24 years with CD19+ B cell malignancies with no available curative treatment options (such as autologous or allogeneic stem cell transplantation) who have a limited prognosis with currently available therapies and were previously treated with a B cell directed engineered cell therapy product.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects with documented CD19+ B cell malignancies and no available curative treatment options (such as autologous or allogeneic SCT) who have limited prognosis (several months to <2 year survival) with currently available therapies will be enrolled:

1. Eligible diseases: CD19+ leukemia or lymphoma. In general, these will be patients with:

   1. ALL without curative options for therapy, including those not eligible for allogeneic SCT. Patient may be in any complete response, or patient may have active disease but responding or stable after most recent therapy.The intent is not to enroll patients with no degree of disease control or rapidly increasing disease burden between enrollment and cell infusion.
   2. Diffuse large cell lymphoma or other high-grade NHL, previously identified as CD19+ including residual disease after primary therapy and not eligible for autologous SCT; relapsed after prior autologous SCT; beyond 1st CR with relapsed or persistent disease and not eligible or appropriate for conventional allogeneic or autologous SCT.
2. Patients previously treated with B cell directed engineered cell therapy are eligible if they meet one of the following criteria:

   1. partial response or no response to prior cell therapy
   2. relapsed after prior cell therapy
   3. demonstrated B cell recovery suggesting loss of engineered cells.
3. Documented CD19 expression (after previous B cell directed cell therapy, if applicable)
4. Age 1 to 24 years
5. Expected survival > 12 weeks
6. Creatinine < 2.5 mg/dl and less than 2.5x normal for age
7. Bilirubin <2.0 mg/dl
8. Adequate pulmonary function defined as < Grade 3 hypoxia
9. Adequate cardiac function defined as LVSF ≥ 28% confirmed by ECHO
10. Adequate performance status (Lansky or Karnofsky score ≥50)
11. Patients with relapsed disease after prior allogeneic SCT (myeloablative or non-myeloablative) will be eligible if they meet all other inclusion criteria and

    1. Have no active GVHD and require no immunosuppression
    2. Are more than 4 months from transplant (6 months at infusion)
12. Patients with CNS3 disease will be eligible if CNS disease is responsive to therapy
13. For those patients who require leukapheresis for T cell collection (i.e. no previously collected product exists), adequate venous access for apheresis or eligible for appropriate catheter placement, and no other contraindications for leukapheresis.
14. Voluntary informed consent is given.

Exclusion Criteria:

1. Pregnant or lactating women. The safety of this therapy on unborn children is not known. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion.
2. Uncontrolled active infection.
3. Active hepatitis B or hepatitis C infection.
4. Concurrent use of systemic steroids at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of physiologic replacement hydrocortisone or inhaled steroids is permitted as well.
5. Presence of grade 2-4 acute or extensive chronic GVHD.
6. Under treatment for GVHD.
7. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity
8. Any uncontrolled active medical disorder that would preclude participation as outlined.
9. HIV infection

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of study related adverse events defined as NCI CTCAE 4.0 > grade 3 possibly, probably, or definitely related to study treatment. | Study treatment until Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Carl June, MD, Study Chair — University of Pennsylvania
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Myers RM, Li Y, Barz Leahy A, Barrett DM, Teachey DT, Callahan C, Fasano CC, Rheingold SR, DiNofia A, Wray L, Aplenc R, Baniewicz D, Liu H, Shaw PA, Pequignot E, Getz KD, Brogdon JL, Fesnak AD, Siegel DL, Davis MM, Bartoszek C, Lacey SF, Hexner EO, Chew A, Wertheim GB, Levine BL, June CH, Grupp SA, Maude SL. Humanized CD19-Targeted Chimeric Antigen Receptor (CAR) T Cells in CAR-Naive and CAR-Exposed Children and Young Adults With Relapsed or Refractory Acute Lymphoblastic Leukemia. J Clin Oncol. 2021 Sep 20;39(27):3044-3055. doi: 10.1200/JCO.20.03458. Epub 2021 Jun 22. PMID 34156874